CLINICAL TRIAL: NCT05044143
Title: Serial Cervical Length Measurements After the 1st Episode of Threatened Preterm Labor to Improve Prediction of Spontaneous Preterm Delivery: Prospective Cohort Study
Brief Title: Prediction of Preterm Delivery with Serial Cervical Length Measurements After Threatened Preterm Labor
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Modena and Reggio Emilia (Other)
Responsible Party: Principal Investigator, Giuseppe Chiossi, Attending Physician, Department of Obstetrics and Gynecology, University of Modena and Reggio Emilia
Other Study IDs: Università di Modena
Record Dates: First submitted 2021-09-03; First posted 2021-09-14 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-01

CONDITIONS: Preterm Labor with Preterm Delivery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Women who remained undelivered after their first episode of threatened preterm labor: Women admitted to the hospital due to their first episode of threatened preterm labor (i.e onset of spontaneous labor < 34 weeks gestation), who did not deliver prematurely as labor stopped (with or without interventions such as tocolysis). Those with a cervical length < 25 mm at the time of hospital discharge are eligible to participate in the study
  Interventions: Other: Monitoring the length of the uterine cervix using transvaginal ultrasound

INTERVENTIONS:
Other: Monitoring the length of the uterine cervix using transvaginal ultrasound — Cervical length is measured with a 7-9 MHz transvaginal probe by trained obstetricians-gynecologists following the same standardized approach (Berghella 2003). Transvaginal CL measurement is largely used in current obstetric practice, and it is considered the 'gold standard' measurement when assessing the uterine cervix. In contrast to transabdominal US, the transvaginal approach is highly reproducible, and measurements are unaffected by maternal obesity, cervical position, and shadowing from fetal parts (Berghella 2003, Hassan 2000, ACOG 2012, Berghella 2012).

SUMMARY:
Prospective cohort study on pregnant women discharged from the hospital after the first episode of threatened preterm labor. Cervical length (CL) will be measured with transvaginal US upon initial presentation (i.e at the time of hospital admission), at the time of hospital discharge, and respectively 2, 4, 8 and 12 weeks later. Pregnant women undelivered after the 1st episode of threatened preterm labor will be invited to participate in the study if CL upon discharge is < 25 mm. The study will investigate the potential association between cervical shortening over time and time of delivery, to assess if spontaneous preterm delivery can be predicted by CL.

DETAILED DESCRIPTION:
Preterm labor is the result of labor occurring prior to 36 6/7 weeks' gestation (i.e spontaneous preterm labor) leading to delivery. Preterm labor is a clinical diagnosis, defined as the appearance of regular contractions accompanied by a change in cervical dilation, effacement, or both, or initial presentation with regular contractions and cervical dilation of at least 2 cm prior to 36 6/7 weeks' gestation.

The pathogenesis of preterm labor has not yet been fully understood, but it has been hypothesized that it could be caused by early idiopathic activation of the normal process of labor or instead, that it could be the result of pathological insults (Goldenberg 2008, Hamilton 2013, Slattery 2002). In Western countries, spontaneous PTB is responsible for 75% of perinatal mortality and more than half of long-term morbidity (McCormick 1985). Although most preterm newborns survive, they have an increased risk of neuro-behavioral disability, cerebral palsy, mental and developmental retardation. Moreover, spontaneous PTB also represents an important cause of chronic broncho pneumopathies, visual and auditory abnormalities and other chronic diseases of the pediatric age including school failure.

As contractions are the most commonly recognized antecedent of preterm birth, cessation of uterine contractions has been the primary focus of therapeutic intervention to prevent the burden of prematurity.

Preterm labor is currently considered a syndrome with a multifactorial etiology, among which inflammation, uteroplacental ischemia or hemorrhage, uterine overdistension, stress and other immune-mediated processes certainly play a role (Romero 2006): these factors do not necessarily represent a direct cause, but contribute to a transition from uterine quiescence to preterm labor or preterm premature rupture of membranes (pPROM) (Goldenberg 2005).

There are many maternal and fetal conditions that have been associated with PTB, including maternal demographic characteristics (such as low socio-economic status, race), nutritional status, obstetric history (history of prior spontaneous PTB), psychological aspects, risk behaviors (such as drug and tobacco use), infections, short CL, as well as biological and genetic markers (Goldenberg 2008, Andrews 2000).

Cervical length is measured with a 7-9 MHz transvaginal probe by trained obstetricians-gynecologists following the same standardized approach (Berghella 2003). Short CL (< 20 mm) prior to 24 weeks' gestation has been recognized as a risk factor for preterm delivery among asymptomatic women; furthermore, short CL (< 25 mm) has also been identified as a risk factor for spontaneous preterm delivery among patients presenting with painful uterine contractions (ACOG 2012).

Threatened preterm labor (TPL) is the most common diagnosis that leads to hospitalization during pregnancy (Bennet 1998) and its annual costs exceed $800 million in the USA (Nicholson 2000). The association between preterm labor and preterm delivery is weak, as less than 10% of women diagnosed preterm labor actually give birth within 7 days of presentation (Fucks 2004). Therefore, clinicians define as threatened preterm labor a condition characterized by uterine contractions associated with cervical changes, that does not lead to preterm delivery, due a spontaneous resolution of the labor process, interventions aimed at possible causes of the labor process (such as treatment of a concomitant infection), or symptomatic therapeutic interventions (such as administration of tocolytics).

Although approximately 75% of women presenting with TPL remain undelivered after a 48-hours course of tocolytics, their risk of preterm delivery remains high, as approximately 30% of them deliver before 37 weeks (Simhan 2007). However, it is a challenge for clinicians to identify who will deliver prematurely after an episode of threatened preterm labor.

Cervical length (CL) measured by transvaginal sonography has been shown to be an accurate predictor of spontaneous preterm delivery among women presenting with painful uterine contractions (Berghella 2017, Sotiriadis 2016). However, studies have mainly focused on the role of a single CL measure collected at the time of the initial presentation instead of evaluating the predictive value of serial CL evaluations as threatened preterm labor resolves. We have previously showed in a secondary analysis of a RCT that serial CL evaluations may help identify those who will deliver prematurely after their first episode of threatened preterm labor (Chiossi 2020). We now intend to validate these findings prospectively, with a cohort study on the role of serial CL measures among women who remained undelivered after their first episode threatened preterm labor. Transvaginal CL measure has the potential to promptly identify shortening of the uterine cervix, a condition associated with preterm delivery. Such evaluation could be included in the antenatal care of women discharged from the hospital after an episode of threatened preterm labor to stratify their risk of preterm birth, to rationalize care and resource-utilization, as well as to improve pregnancy outcome.

Pregnant women admitted to the hospital with the diagnosis of threatened preterm labor (regular contractions accompanied a change in cervical dilation, effacement, or both, or initial presentation with regular contractions and cervical dilation of at least 2 cm), who remained undelivered, will be invited to participate if CL upon discharge is < 25 mm. Cervical length will be evaluated at follow up appointments 2, 4, 8 and 12 weeks after discharge and linked to the actual gestational age at delivery.

Using a CL threshold of 10 mm we will estimate the risk of preterm delivery at different time points: each risk assessment will be based on the CL measured from hospital admission up to that time. At hospital discharge, patients will be classified at "low risk" of preterm delivery if their CL will be > 10 mm, while "high risk" subjects will have a shorter CL. The risk of preterm birth will then be assessed on all the women who will remain undelivered until the 1st follow up appointment, 2 weeks later: pregnancies with CL measurements > 10 mm from hospital discharge up to 2 weeks later will be considered "low risk", while those with CL < 10 mm on at least one assessment will be classified as "high risk". If delivery will not occur after 4 weeks (2nd follow up visit), pregnancies who will maintain CL measurement > 10 mm from hospital admission through the following 2 visits will be classified as "low risk", while "high risk" women will have a shorter CL on at least one of the 4 assessments. Risk estimates will be calculated in a similar fashion on women still pregnant 8 and 12 weeks after hospital discharge (3rd and 4th follow up visits). Cervical length will also be evaluated upon hospital admission, and the risk of preterm delivery will also be assessed taking into account such value.

Descriptive statistics will be used to characterize the socio-demographic features and the obstetric characteristics of women categorized as "low risk" (i.e pregnancies whose CL persistently remains above 10 mm) or high risk (i.e those with at least one CL measurement < 10 mm): categorical variables will be presented as absolute and percentage frequencies, they will be tested with Chi square test or Fisher's exact test as appropriate. Continuous variables will be summarized as mean +/- SD and compared with Student's t test. A level of statistical significance of p < 0.05 will be considered.

To control for confounding, multivariate logistic regression models will be used to describe the association between delivery prior to 37 weeks' gestation and CL (measured from hospital admission to each subsequent evaluation). Socio-demographic variables such as maternal age, BMI at entry to care, ethnicity, smoking, and education will be considered as potential confounders. Similarly, obstetric features such as parity, tocolysis at the initial hospitalization or at any subsequent hospital admission, urine culture collected on the initial hospitalization, and gestational age at enrolment will also be tested as potential.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy at 23+0 - 33+6 weeks' gestation
* Age > 18 years old
* Patients should be capable of providing consent to participate in the study

Exclusion Criteria:

* Previous spontaneous preterm (20+0 - 36+6 weeks' gestation) delivery (including history of pregnancy loss due to cervical incompetence, i.e painless cervical dilatation prior to 24 weeks' gestation)
* Treatment with 17 hydroxyprogesterone caproate due to a previous spontaneous preterm delivery
* Detection of a cervical length < 25 mm during routine ultrasound < 24 weeks' gestation in asymptomatic patients (i.e patients that do not complain of uterine contractions or patients with no uterine contractions documented on tocometry)
* Treatment with vaginal progesterone or micronized progesterone due to a cervical length < 25 mm
* Cerclace placement in the current or in a previous pregnancy
* Multiple pregnancy
* Age < 18 years old
* Preterm premature rupture of membranes (pPROM) upon initial presentation
* Müllerian malformations
* Prior cervical surgery

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — The study will be conducted on pregnant women
Study Population: Women who remained undelivered after their first episode of threatened preterm labor, whose cervical length upon hospital discharge is < 25 mm
Sampling Method: Non-Probability Sample
Enrollment: 303 (Estimated)
Dates: Start 2021-10-20 (Actual); Primary Completion 2025-06-20 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
To investigate the association between cervical length measured at different time points and the risk of spontaneous preterm birth < 37 weeks' gestation | At the time of delivery
  The risk of spontaneous preterm birth < 37 weeks' gestation will be compared among women with at least a cervical length < 10 mm as opposed to those whose cervix will remain persistently > 10 mm. A relationship between gestational age at delivery and cervical length will also be investigate considering the two variables as continuous

SECONDARY OUTCOMES:
To assess a possible association between cervical length and adverse neonatal outcomes | At the time of delivery
  Adverse neonatal outcomes will be summarized as a composite of neonatal death, neonatal resuscitation, non-invasive (cPAP) or invasive (mechanical ventilation) respiratory support, hypoglycemia (< 44 mg/dl needing therapy), newborn sepsis, confirmed seizures, stroke, intraventricular hemorrhage (IVH), basal nuclei anomalies, cardiopulmonary resuscitation, umbilical-cord-blood arterial pH < 7.0 or base excess < -12.5, prolonged hospitalization (> 5 days), or shoulder dystocia.
To assess a possible association between cervical length and adverse maternal outcomes. | At the time of delivery
  Adverse maternal outcomes will be summarized as a composite of blood loss > 1000 ml, maternal sepsis, post-partum endometritis, hysterectomy, bowel or urinary tract injuries, uterine rupture, wound (either perineal or abdominal) complications (i.e abscess, hematoma or disruption), 3rd and 4th degree perineal lacerations, blood transfusion, maternal admission to the ICU, laparotomy, and death.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Chiossi, MD, Principal Investigator — Dept of Ob/Gyn, Modena Policlinico Hospital, University of Modena and Reggio Emilia
Locations (6):
- Italy (6):
  - Facoltà di Medicina e Chirurgia, università politecnica delle Marche, Ancona
  - Mariarosaria Di Tommaso, Divisione di Ginecologia ed Ostetricia, Dipartimento Assistenziale Integrato Materno Infantile, Azienda Ospedaliero-Universitaria Careggi, Florence
  - Divisione di Ginecolgia ed stetricia, Azienda Ospedaliera Vimercate-Desio presidio di Carate Brianza Giussano, e Università di Milano Bicocca, Milan
  - Fondazione IRCCS Cà Granda, Ospedale Maggiore Policlinico, Clinica Mangiagalli, Università di Milano, Milan
  - Department of Obstetrics and Gynecology, Foundation MBBM at San Gerardo Hospital, University of Milan-Bicocca School of Medicine and Surgery, Monza
  - Divisione di Ginecologia ed Ostetricia, Dipartimento Materno infantile, Arcispedale Santa Maria Nuova, IRCCS, Reggio Emilia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andrews WW, Copper R, Hauth JC, Goldenberg RL, Neely C, Dubard M. Second-trimester cervical ultrasound: associations with increased risk for recurrent early spontaneous delivery. Obstet Gynecol. 2000 Feb;95(2):222-6. doi: 10.1016/s0029-7844(99)00483-4. PMID 10674583
- [Background] Bennett TA, Kotelchuck M, Cox CE, Tucker MJ, Nadeau DA. Pregnancy-associated hospitalizations in the United States in 1991 and 1992: a comprehensive view of maternal morbidity. Am J Obstet Gynecol. 1998 Feb;178(2):346-54. doi: 10.1016/s0002-9378(98)80024-0. PMID 9500498
- [Background] Berghella V, Bega G, Tolosa JE, Berghella M. Ultrasound assessment of the cervix. Clin Obstet Gynecol. 2003 Dec;46(4):947-62. doi: 10.1097/00003081-200312000-00026. No abstract available. PMID 14595237
- [Background] Berghella V, Palacio M, Ness A, Alfirevic Z, Nicolaides KH, Saccone G. Cervical length screening for prevention of preterm birth in singleton pregnancy with threatened preterm labor: systematic review and meta-analysis of randomized controlled trials using individual patient-level data. Ultrasound Obstet Gynecol. 2017 Mar;49(3):322-329. doi: 10.1002/uog.17388. Epub 2017 Feb 8. PMID 27997053
- [Background] Society for Maternal-Fetal Medicine Publications Committee, with assistance of Vincenzo Berghella. Progesterone and preterm birth prevention: translating clinical trials data into clinical practice. Am J Obstet Gynecol. 2012 May;206(5):376-86. doi: 10.1016/j.ajog.2012.03.010. PMID 22542113
- [Background] Chiossi G, Facchinetti F, Vergani P, Di Tommaso M, Marozio L, Acaia B, Pignatti L, Locatelli A, Spitaleri M, Benedetto C, Zaina B, D'Amico R; PROTECT Collaborative Group. Serial cervical-length measurements after first episode of threatened preterm labor improve prediction of spontaneous delivery prior to 37 weeks' gestation. Ultrasound Obstet Gynecol. 2021 Feb;57(2):298-304. doi: 10.1002/uog.22188. PMID 32851714
- [Background] Committee on Practice Bulletins-Obstetrics, The American College of Obstetricians and Gynecologists. Practice bulletin no. 130: prediction and prevention of preterm birth. Obstet Gynecol. 2012 Oct;120(4):964-73. doi: 10.1097/AOG.0b013e3182723b1b. No abstract available. PMID 22996126
- [Background] Friedman AM, Schwartz N, Ludmir J, Parry S, Bastek JA, Sehdev HM. Can transabdominal ultrasound identify women at high risk for short cervical length? Acta Obstet Gynecol Scand. 2013 Jun;92(6):637-41. doi: 10.1111/aogs.12111. Epub 2013 Apr 17. PMID 23590553
- [Background] Fuchs IB, Henrich W, Osthues K, Dudenhausen JW. Sonographic cervical length in singleton pregnancies with intact membranes presenting with threatened preterm labor. Ultrasound Obstet Gynecol. 2004 Oct;24(5):554-7. doi: 10.1002/uog.1714. PMID 15386604
- [Background] Goldenberg RL, Culhane JF, Iams JD, Romero R. Epidemiology and causes of preterm birth. Lancet. 2008 Jan 5;371(9606):75-84. doi: 10.1016/S0140-6736(08)60074-4. PMID 18177778
- [Background] Goldenberg RL, Culhane JF. Prepregnancy health status and the risk of preterm delivery. Arch Pediatr Adolesc Med. 2005 Jan;159(1):89-90. doi: 10.1001/archpedi.159.1.89. No abstract available. PMID 15630064
- [Background] Gomez R, Romero R, Medina L, Nien JK, Chaiworapongsa T, Carstens M, Gonzalez R, Espinoza J, Iams JD, Edwin S, Rojas I. Cervicovaginal fibronectin improves the prediction of preterm delivery based on sonographic cervical length in patients with preterm uterine contractions and intact membranes. Am J Obstet Gynecol. 2005 Feb;192(2):350-9. doi: 10.1016/j.ajog.2004.09.034. PMID 15695971
- [Background] Hamilton BE, Martin JA, Ventura SJ. Births: preliminary data for 2012. Natl Vital Stat Rep. 2013 Sep;62(3):1-20. PMID 24321416
- [Background] Hassan SS, Romero R, Berry SM, Dang K, Blackwell SC, Treadwell MC, Wolfe HM. Patients with an ultrasonographic cervical length < or =15 mm have nearly a 50% risk of early spontaneous preterm delivery. Am J Obstet Gynecol. 2000 Jun;182(6):1458-67. doi: 10.1067/mob.2000.106851. PMID 10871466
- [Background] Hernandez-Andrade E, Romero R, Ahn H, Hussein Y, Yeo L, Korzeniewski SJ, Chaiworapongsa T, Hassan SS. Transabdominal evaluation of uterine cervical length during pregnancy fails to identify a substantial number of women with a short cervix. J Matern Fetal Neonatal Med. 2012 Sep;25(9):1682-9. doi: 10.3109/14767058.2012.657278. Epub 2012 Mar 16. PMID 22273078
- [Background] Honest H, Bachmann LM, Gupta JK, Kleijnen J, Khan KS. Accuracy of cervicovaginal fetal fibronectin test in predicting risk of spontaneous preterm birth: systematic review. BMJ. 2002 Aug 10;325(7359):301. doi: 10.1136/bmj.325.7359.301. PMID 12169504
- [Background] McCormick MC. The contribution of low birth weight to infant mortality and childhood morbidity. N Engl J Med. 1985 Jan 10;312(2):82-90. doi: 10.1056/NEJM198501103120204. PMID 3880598
- [Background] Nicholson WK, Frick KD, Powe NR. Economic burden of hospitalizations for preterm labor in the United States. Obstet Gynecol. 2000 Jul;96(1):95-101. doi: 10.1016/s0029-7844(00)00863-2. PMID 10862850
- [Background] Owen J, Iams JD; National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. What we have learned about cervical ultrasound. Semin Perinatol. 2003 Jun;27(3):194-203. doi: 10.1016/s0146-0005(03)00021-1. PMID 12889586
- [Background] Romero R, Espinoza J, Kusanovic JP, Gotsch F, Hassan S, Erez O, Chaiworapongsa T, Mazor M. The preterm parturition syndrome. BJOG. 2006 Dec;113 Suppl 3(Suppl 3):17-42. doi: 10.1111/j.1471-0528.2006.01120.x. PMID 17206962
- [Background] Saigal S, Doyle LW. An overview of mortality and sequelae of preterm birth from infancy to adulthood. Lancet. 2008 Jan 19;371(9608):261-9. doi: 10.1016/S0140-6736(08)60136-1. PMID 18207020
- [Background] Simhan HN, Caritis SN. Prevention of preterm delivery. N Engl J Med. 2007 Aug 2;357(5):477-87. doi: 10.1056/NEJMra050435. No abstract available. PMID 17671256
- [Background] Slattery MM, Morrison JJ. Preterm delivery. Lancet. 2002 Nov 9;360(9344):1489-97. doi: 10.1016/S0140-6736(02)11476-0. PMID 12433531
- [Background] Sonek JD, Iams JD, Blumenfeld M, Johnson F, Landon M, Gabbe S. Measurement of cervical length in pregnancy: comparison between vaginal ultrasonography and digital examination. Obstet Gynecol. 1990 Aug;76(2):172-5. PMID 2196494
- [Background] Sotiriadis A, Papatheodorou S, Kavvadias A, Makrydimas G. Transvaginal cervical length measurement for prediction of preterm birth in women with threatened preterm labor: a meta-analysis. Ultrasound Obstet Gynecol. 2010 Jan;35(1):54-64. doi: 10.1002/uog.7457. PMID 20014326